CLINICAL TRIAL: NCT02962583
Title: The Addition of Probiotic Consumption to a Nutritional Intervention and Caloric Restriction on Body Weight and Composition in Overweight Participants: A Randomized, Double-blind, Placebo Controlled Study
Brief Title: The Addition of Probiotic Consumption to a Nutritional Intervention and Caloric Restriction on Body Weight and Composition in Overweight Participants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Lallemand Health Solutions (Industry)
Responsible Party: Principal Investigator, Angelo Tremblay, Professor, Laval University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLIN-21-012
Record Dates: First submitted 2016-11-02; First posted 2016-11-11 (Estimated); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Probiotic (Experimental): Daily probiotic consumption
  Interventions: Other: Weight loss; Drug: Probiotic Formula
- Placebo (Placebo Comparator): Daily placebo consumption
  Interventions: Other: Weight loss; Drug: Placebos

INTERVENTIONS:
Other: Weight loss
Drug: Probiotic Formula
  Arms: Probiotic
Drug: Placebos
  Arms: Placebo

SUMMARY:
Limited interventional human studies suggest that probiotic supplementation may be a beneficial strategy for promoting weight loss when added to a nutritional intervention via their effects on lipid absorption and metabolic signaling molecules. The purpose of this study is to evaluate the effects of addition of a probiotic supplementation to a weight loss intervention on body weight, body composition and overall health in overweight adults.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 55 years
* BMI between 27.0 and 39.9 kg/m2
* Sedentary to moderate active (less than 30 minutes of physical activity, 3 times per week)
* Willingness to complete questionnaires, records, and diaries associated with the study and to complete all study visits
* Willingness to discontinue consumption of fermented foods or probiotics (e.g. yoghourts, with live, active cultures or supplements), laxatives, prebiotics and any substance for body weight control
* Willingness and ability to provide informed consent in French
* Willingness to receive random assignment to probiotic or placebo supplementation
* Committed to losing weight over the 12-week study period

Exclusion Criteria:

* Smokers
* Use of another investigational product within three months of the pre-baseline period.
* Known to be pregnant or breast-feeding or planning on becoming pregnant in the next 18 months.

  * Women of child-bearing potential not using effective contraception which include:
  * Hormonal contraceptives including combined oral contraceptives, hormone birth control patch, vaginal contraceptive ring, injectable contraceptives, or hormonal implants
  * Intrauterine devices (IUD) or Intrauterine system (IUS)
  * Tubal ligation
  * Vasectomy of partner
  * Double barrier method (use of physical barrier by both partners, e.g. male condom and diaphragm, male condom and cervical cap)
* Positive pregnancy test in women of child-bearing potential
* Menopausal women
* Allergic to milk, soy, or yeast
* Weight gain or loss of at least 10 lbs in previous three months
* Inflammatory bowel syndrome, celiac disease, short bowel syndrome, or any other malabsorptive syndrome
* Uncontrolled angina within the past six months
* Insulin-dependent diabetes (oral medications are not exclusionary)
* Serious and/or unstable medical conditions (e.g. cardiovascular, renal, lung, psychiatric illness, bleeding disorders, etc.)
* Cancer treatment (radiation, chemotherapy, surgery) within past six months or any other treatment or condition known to weaken the immune system (such as systemic corticosteroids or HIVIAIDS).
* Any physical condition deemed likely to significantly interfere with individuals' ability to participate in a nutritional intervention.
* Currently or at any point during the study participating in Weight Watcher's or another weight loss program or taking a medication for weight loss.
* Under antibiotics or treatments (medication or nutritional program) affecting body weight Intake and/or energy expenditure
* History of drug or alcohol (> 9 drinks weekly) abuse
* Abnormal thyroid hormone levels
* Immune-compromised conditions
* Participant experiencing nausea, fever, vomiting, bloody diarrhoea or severe abdominal pain

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 152 (Actual)
Dates: Start 2017-01; Primary Completion 2019-06-06 (Actual); Study Completion 2019-06-06 (Actual)

PRIMARY OUTCOMES:
Change from Baseline body weight at 12 weeks | 12 weeks

SECONDARY OUTCOMES:
Change from Baseline BMI at 12 weeks | 12 weeks
Change from Baseline waist circumference data at 12 weeks | 12 weeks
Change from Baseline sagittal abdominal diameter data at 12 weeks | 12 weeks
Change from Baseline body composition at 12 weeks | 12 weeks
  DXA
Change from Baseline stress level at 12 weeks | 12 weeks
  Questionnaire
Change from Baseline anxiety level at 12 weeks | 12 weeks
  Questionnaire
Change from Baseline depression symptoms at 12 weeks | 12 weeks
  Questionnaire
Change from Baseline sleeping habits at 12 weeks | 12 weeks
  Questionnaire
Change from Baseline intestinal microbiota composition at 12 weeks | 12 weeks
  Changes in the concentrations of the probiotic strains in the stools will be measured with strain specific DNA in fecal samples.
Change from Baseline C-reactive protein at 12 weeks | 12 weeks
Change from Baseline TNF-a at 12 weeks | 12 weeks
Change from Baseline interleukin-6 at 12 weeks | 12 weeks
Change from Baseline lipopolysaccharide (LPS) at 12 weeks | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Angelo Tremblay, Ph.D, Study Director — Laval University
Locations (1):
- PEPS - Université Laval, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Choi BS, Brunelle L, Pilon G, Cautela BG, Tompkins TA, Drapeau V, Marette A, Tremblay A. Lacticaseibacillus rhamnosus HA-114 improves eating behaviors and mood-related factors in adults with overweight during weight loss: a randomized controlled trial. Nutr Neurosci. 2023 Jul;26(7):667-679. doi: 10.1080/1028415X.2022.2081288. Epub 2022 Jun 17. PMID 35714163